CLINICAL TRIAL: NCT02924662
Title: The Investigation of the Depression in Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dalian Municipal Central Hospital (Other)
Responsible Party: Principal Investigator, Wenjun Wang, MD, Dalian Municipal Central Hospital
Other Study IDs: DaLianMCH
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Kellgren and Lawrence classification I: Grade I Kellgren and Lawrence radiographic changes.
  Interventions: Other: There is no intervention.
- Kellgren and Lawrence classification II: Grade II Kellgren and Lawrence radiographic changes.
- Kellgren and Lawrence classification III: Grade III Kellgren and Lawrence radiographic changes.
- Kellgren and Lawrence classification IV: Grade IV Kellgren and Lawrence radiographic changes.

INTERVENTIONS:
Other: There is no intervention.
  Groups: Kellgren and Lawrence classification I

SUMMARY:
Studies have reported that the patient's psychological state such as anxiety, depression and other emotion affect the therapeutic effect of osteoarthritis, also may be the important reason for the poor knee joint osteoarthritis efficacy.

The aim of this study are firstly to investigate the depression status of patients with osteoarthritis. Secondly, the study will aim to assess whether osteoarthritis progression will affect depression status, ultimately, provide reference for clinical.

ELIGIBILITY:
Inclusion Criteria:

Meet the 1986 American College of Rheumatology (ACR) clinical criteria for knee osteoarthritis and the 2010 Chinese Medical Association clinical criteria for knee osteoarthritis.

Exclusion Criteria:

Patients with rheumatoid arthritis patients with a history of depression before osteoarthritis pathogenesis patients who can't cooperate with related inspection and assessment Patients with mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will be taken from a single centre. The patient population will be patients who are diagnosed with osteoarthritis. Participants will have a comprehensive and detailed assessment by a qualified doctor. After the assessment，the participants who are diagnosed with osteoarthritis and conformed to fit the eligibility criteria will be invited to join the investigation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster OA index (WOMAC) | Day 1
American knee society knee score | Day 1
Hamilton Depression Scale-17（HAMD-17） | Day 1